CLINICAL TRIAL: NCT05172323
Title: Pre-procedural 3D Reconstructed Computer Tomography Versus Angiography Guided Percutaneous Coronary Intervention for Ostial Right Coronary Artery Lesions
Brief Title: Pre-procedural 3DCT Versus Angiography Guided PCI for Ostial Right Coronary Artery Lesions
Acronym: 3DCT-RCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Koen Ameloot, Interventional cardiologist, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z-2021107
Record Dates: First submitted 2021-11-24; First posted 2021-12-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: Right coronary artery; Computed tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: A prospective, investigator-initiated, single-centre, randomized-controlled, assessor blinded pilot trial.
Who Masked: Outcomes Assessor
Masking Description: The assessor of the IVUS images will be blinded to treatment arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3DCT-guided group (Experimental): PCI guided with 3DCT results and IVUS
  Interventions: Device: 3DCT-scan
- Angiography-guided group (Placebo Comparator): PCI guided by operator and IVUS
  Interventions: Other: Angiography guided PCI

INTERVENTIONS:
Device: 3DCT-scan — A contrast CT-scan of the coronary arteries will be performed and 3D analyzed to determine the best angle for the C-arm during Percutaneous Coronary Intervention (PCI) for stent implantation. Furthermore determining the amount and localization of calcium in the right coronary artery (RCA) and diameter and length of RCA. The use of IVUS will be used to determine the degree of calcium.
  Arms: 3DCT-guided group
Other: Angiography guided PCI — Standard of care is angiography guided PCI of the ostium of the RCA. The use of IVUS will be used to determine the degree of calcium.
  Arms: Angiography-guided group

SUMMARY:
Even with second generation drug eluting stents, rates of target lesion failure (TLF) for aorto-ostial RCA lesions remain high [3yrs TLF 14.2%]. Retrospective studies show that stent underexpansion and geographical stent-ostium mismatch are the main predictors for TLF. Geographical mismatch means that the stent is implanted either too distal (thereby not fully covering the lesion) or too proximal (thereby protruding too much in the aorta and hampering future engagement with guiding catheters). The investigators hypothesize that, pre-procedural 3D CT coronarography to determine the optimal C-arm angle of the X-ray system with the most accurate visualization of the aorto-ostial angle and determination of localization of calcium, could prevent geographical mismatch.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated non-emergent PCI for an aorta-ostial-RCA lesion defined as a significant de novo lesion [by angiography or by physiological assessment] for which the operator intends to fully cover the ostial RCA with stent struts
* Willing to provide informed consent

Exclusion Criteria:

* Emergent PCI indication: if the ostial RCA lesion is the culprit lesion of an acute coronary syndrome [of note: if the ostial RCA lesion is a non-culprit lesion, patient can be included in the trial]
* In-stent restenosis or thrombosis in the ostial RCA
* Renal insufficiency [eGFR<30 ml/min]
* Known allergic reaction to contrast medium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Geographical mismatch as quantified by intra-coronary ultrasound (IVUS) | Procedural
  Distance between the aorta-ostial junction and the most proximal protruding stent strut (in mm).

SECONDARY OUTCOMES:
Geographical mismatch as quantified by intra-coronary ultrasound (IVUS) | Procedural
  Percentage of patients without geographical mismatch as defined by a fully covered ostium AND a maximal length between the aorta-ostial junction and the most proximal protruding stent struts not more then 3mm
Geographical mismatch as quantified by intra-coronary ultrasound (IVUS) | Procedural
  The percentage of patients who need an additional stent after the final IVUS has shown that the ostium was not fully covered
Volume of contrast agent administered | Procedural
  Expressed in mL
Procedural radiation dose | Procedural
  Expressed in mGy
Procedural duration from first puncture of artery to skin closure | Procedural
  Expressed in minutes
Minimal luminal area (MLA) | Procedural
  The predicted MLA by 3DCT will be compared with the MLA prior to stent placement as obtained with IVUS
Stent sizing | Procedural
  Predicted stent diameter and length by 3DCT will be compared with the effectively implanted stent size
Stent expansion | Procedural
  Expressed as the minimal stent area (MSA) determined by IVUS, divided by the reference luminal area in the healthy distal landing zone
Calcium modification | Procedural
  Prediction of calcium modification pre-IVUS compared with IVUS based strategy of calcium modification
Calcified lesions | Procedural
  Calcium score as determined by 3DCT will be correlated with the maximum calcium arc on IVUS
MACCE at 30 days follow-up | 30 days after PCI
  30 days event rate [death, non-fatal MI, non-fatal stroke, definite or probable stent thrombosis, target lesion failure]

CONTACTS AND LOCATIONS:
Overall Officials: Koen Ameloot, Dr., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Background] Mitomo S, Jabbour RJ, Watanabe Y, Mangieri A, Ancona M, Regazzoli D, Tanaka A, Nakajima A, Naganuma T, Giannini F, Latib A, Nakamura S, Colombo A. Comparison of mid-term clinical outcomes after treatment of ostial right coronary artery lesions with early and new generation drug-eluting stents: Insights from an international multicenter registry. Int J Cardiol. 2018 Mar 1;254:53-58. doi: 10.1016/j.ijcard.2017.10.066. Epub 2018 Jan 28. PMID 29407132
- [Derived] van den Buijs DMF, Poels EM, Willems E, Cottens D, Dotremont K, De Leener K, Meekers E, Ferdinande B, Vrolix M, Dens J, Ameloot K. Three-Dimensional CT for Preprocedural Planning of PCI for Ostial Right Coronary Artery Lesions: A Randomized Controlled Pilot Trial. Circ Cardiovasc Interv. 2025 Feb;18(2):e013584. doi: 10.1161/CIRCINTERVENTIONS.123.013584. Epub 2025 Jan 29. PMID 39878016